CLINICAL TRIAL: NCT02429674
Title: The Efficacy of a Depression Intervention for Adolescents With Depression and Sleep Disturbances
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Principal Investigator, Eleanor McGlinchey, Assistant Professor of Clinical Psychology in Psychiatry, New York State Psychiatric Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: #7089
Record Dates: First submitted 2015-04-22; First posted 2015-04-29 (Estimated); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Depression
Keywords: Depression; Adolescence
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TranS-C and IPT-A (Other): 12 sessions of weekly outpatient psychotherapy for adolescent depression.
  Interventions: Behavioral: TranS-C and IPT-A

INTERVENTIONS:
Behavioral: TranS-C and IPT-A — The goal of IPT-A is to decrease depressive symptoms by focusing on current interpersonal difficulties and helping the adolescent improve his or her relationships and interpersonal interactions. This is accomplished through psychoeducation about the adolescent's depression and its link to interpersonal relationships, review of the adolescent's significant relationships, identification of interpersonal problem areas on which to focus the treatment, development of interpersonal problem solving and communication skills, and role-playing. The sleep disturbances intervention will include several modules selected because they are successful treatments for insomnia, and/or may help promote adherence to some of the recommendations related to sleep.
  Other Names: Transdiagnostic Sleep and Circadian treatment and IPT-A

SUMMARY:
The focus of this study is on identifying how Interpersonal Psychotherapy for Adolescents (IPT-A) with depression works to change sleep and related biological markers found in saliva, namely cortisol and pro-inflammatory cytokine levels. The long-term goal of this project is to understand the biological mechanisms of recovery from depression in order to assist in selecting and guiding personalized psychotherapeutic interventions with the highest likelihood of success for individual adolescents with depression.

DETAILED DESCRIPTION:
The primary aim of this project is to examine whether adolescent depression and the associated symptoms of sleep disturbance are best treated using an empirically supported psychotherapy that is augmented with a sleep improvement module. Twenty adolescents (ages 12-17) who meet criteria for major depressive disorder, dysthymic disorder, depressive disorder not otherwise specified, or adjustment disorder with depressed mood and also report elevated levels of sleep disturbance will receive Interpersonal Psychotherapy for Depressed Adolescents (IPT-A) with an adjunctive sleep module that is integrated throughout the treatment. Identifying the best approach to treating both the adolescent's depression and the commonly associated symptom of sleep disturbance will have significant implications for the long-term outcomes of depressed adolescents. Moreover, identifying unique symptom and biological profiles at the outset of treatment may enable doctors to predict treatment outcome.

ELIGIBILITY:
Inclusion Criteria:

* outpatient participant
* parent or legally authorized representative must provide consent and assent by the participant
* Diagnostic and Statistical Manual of Mental Disorders Fifth Edition (DSM-V) criteria for a depressive disorder
* Clinical Global Assessment Scale (C-GAS) < 65
* Quick Inventory of Depression Symptoms - Self Report 16 (QIDS-SR16) over 8 and less than 24.
* English speaking
* significant sleep complaints

Exclusion Criteria:

* co-morbid psychiatric diagnosis of bipolar disorder, psychosis, autism spectrum disorder, intellectual development disorder, conduct disorder or substance abuse disorder
* any condition or illness such as uncontrolled seizure disorder, uncontrolled diabetes, or any other conditions that represent as an inappropriate risk to the participant and/or could confound the interpretation of the study
* currently in active evidence-based psychotherapy for the same condition
* currently taking medication for a psychiatric diagnosis that is not a stable dose (4 weeks on the same dose).
* currently considered at risk for suicide in the opinion of the study doctor, has made a suicide attempt in the past 4 months, or is currently reporting active suicidal ideation.
* history of alcohol or other substance abuse as defined by DSM-V within the last 6 months.
* evidence from clinical diagnosis or report by youth or parent of sleep apnea, restless legs or periodic limb movements during sleep
* sleep treatment that might confound the interpretation of sleep outcomes.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 14 (Actual)
Dates: Start 2015-02; Primary Completion 2020-10 (Actual); Study Completion 2021-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Depression symptom score on the Children's Depression Rating Scale (CDRS) | Week 12
  Reduction in depression symptoms

SECONDARY OUTCOMES:
Change from Baseline in sleep using actigraphy estimated sleep variables | Week 12
  Reduction in sleep difficulties and increase in sleep duration
Change from baseline in Cytokine levels found in saliva | Week 12
  Reduction in inflammatory markers

CONTACTS AND LOCATIONS:
Overall Officials: Eleanor L McGlinchey, Ph.D., Principal Investigator — New York State Psychiatric Institute
Locations (1):
- Pediatric Anxiety and Mood Research Clinic, New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No